CLINICAL TRIAL: NCT03959683
Title: A Prospective Randomized Multicenter Trial Comparing Performance of Two Intracorporeal Lithotripters for Removal of Large Renal Calculi
Brief Title: ShockPulse-SE vs. Trilogy Trial: Comparing the Performance of Two Intracorporeal Lithotripters for Removal of Large Renal Calculi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Boston Scientific Corporation (Industry); Ohio State University (Other); Mayo Clinic (Other); University of British Columbia (Other)
Responsible Party: Principal Investigator, Tim Large, Assistant Professor Urology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1803658961
Record Dates: First submitted 2019-05-16; First posted 2019-05-22 (Actual); Results first posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Kidney Calculi
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, multicenter, 2 arm, comparative trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Trilogy device (Active Comparator): Trilogy Lithotrite to fragment urinary tract calculi in the kidney, ureter and bladder
  Interventions: Device: Trilogy Lithotrite
- ShockPulse-SE (Active Comparator): ShockPulse-SE Lithotripsy System to fragment urinary calculi in the kidney, ureter and bladder
  Interventions: Device: The ShockPulse-SE Lithotripsy System

INTERVENTIONS:
Device: Trilogy Lithotrite — The Trilogy has been FDA cleared for fragmentation of urinary tract calculi in the kidney, ureter, and bladder. Trilogy is a combined piezoelectric/pneumatic device capable of fragmenting calculi and aspirating stone debris. The novel technology in Trilogy has been demonstrated in bench testing to more quickly disintegrate stones compared to other devices.
  Arms: Trilogy device
Device: The ShockPulse-SE Lithotripsy System — The ShockPulse-SE System is an electromechanical device capable of fragmenting calculi and aspirating stone debris. The novel technology in the ShockPulse-SE Lithotripsy System uses a single transducer and proprietary ShockPulse technology to generate both low-frequency mechanical impacts and high-frequency ultrasonic energy which quickly disintegrates stones.
  Arms: ShockPulse-SE

SUMMARY:
The purpose of this study is to measure how well two different devices work to break up and remove kidney stones. We are comparing a newer device to an older one to see which one is faster at breaking up kidney stones. We hypothesize that the Trilogy will increase the stone clearance rate by 25% compared to the Shockpulse-SE

DETAILED DESCRIPTION:
Large and complex renal calculi, defined as those with a maximum diameter of ≥ 1.5 cm, can be removed from the upper urinary tract by percutaneous nephrolithotomy but the stones usually require fragmentation in order to remove them through the access site. There are a number of commercially available intracorporeal lithotripters used to fragment or break kidney stones to allow elimination including pneumatic, ultrasonic, and combination devices. Each technology has its own relative advantages and disadvantages.

New versions of intracorporeal lithotripter devices have been introduced with improvements meant to address prior functional limitations such as probe clogging or breaking and cumbersome hand piece design.

The Trilogy lithotrite is the newest generation device stone fragmentation device from Boston Scientific. The Trilogy device uses unique technology to efficiently fragment and remove stone material, superior to other devices on the market based on preliminary bench testing. From Olympus, the ShockPulse-SE Lithotripsy System (Cybersonics, Erie, PA, USA) is a constant ultrasonic wave energy lithotripter with intermittent shock wave (ballistic/mechanical) energy. The ShockPulse-SE has a single probe design with an OD of 3.76 mm which allows for larger sized stone fragments to be vacuumed from the urothelium. The larger, single lumen also allows for a high flow rate to reduce probe clogging events. The end result is faster stone clearance rates based on in vitro studies.

The objective of this study is to compare the performance, as measured by the stone clearance rate at time of percutaneous nephrolithotomy, of the ShockPulse-SE Lithotripsy System to the Trilogy lithotrite when used for large complex renal calculi.

The Trilogy has been FDA cleared for fragmentation of urinary tract calculi in the kidney, ureter, and bladder. Trilogy is a combined piezoelectric/pneumatic device capable of fragmenting calculi and aspirating stone debris. The novel technology in Trilogy has been demonstrated in bench testing to more quickly disintegrate stones compared to other devices.

The ShockPulse-SE Lithotripsy System has been FDA cleared fragmentation of urinary tract calculi in the kidney, ureter, and bladder. The ShockPulse-SE System is an electromechanical device capable of fragmenting calculi and aspirating stone debris. The novel technology in the ShockPulse-SE Lithotripsy System uses a single transducer and proprietary ShockPulse technology to generate both low-frequency mechanical impacts and high-frequency ultrasonic energy which quickly disintegrates stones.

Study Objectives To compare the performance, as measured by the stone clearance rate at time of percutaneous nephrolithotomy, of the ShockPulse-SE Lithotripsy System to the Trilogy Lithotrite.

Study Endpoints Primary Endpoint Stone clearance rate defined as the kidney stone surface area measured by preoperative computed tomography (CT) scan divided by the time to remove the targeted stone burden.

Time to remove the targeted stone burden is measured at time the lithotripter unit starts fragmenting the stone to time all fragments are removed from the kidney based on visual inspection. This is prior to final visual inspection of the kidney with a flexible nephroscope.

Additional Endpoints

1. Device malfunctions
2. All complications measured by the Clavien Classification of Surgical Complications Stone free status as defined by the presence or absence of stone material on postoperative day 1 CT imaging This study is a post-market, prospective, randomized, multicenter, 2-arm, comparative trial.

Scale and Duration A total of 100 participants will be enrolled and treated at 4 study sites (3 USA, 1 Canada). Two sites will enroll 16 participants and 2 will enroll at least 18 participants. Each subject will be followed for approximately 6-12 weeks after the study procedure. It is anticipated for the entire study to last approximately 12 months.

Treatment Assignment The participants will be block randomized 1:1 to either stone removal with the Trilogy or the ShockPulse-SE device. All randomization will occur at the central study site via computer randomization by the statistician to limit selection bias.

Justification for the Study Design This study will compare performance of two devices for the treatment of large renal calculi. The study has been designed as a prospective, multi-centric, randomized, comparative study. The intent of this design is to minimize bias and to allow for statistical comparison of the two treatment groups.

Point of Enrollment A participant will be considered enrolled in the study if they meet all eligibility criteria and after the participant signs and dates the informed consent form (ICF). No study-related procedures can take placed until the ICF is signed.

Withdrawal All participants enrolled in the clinical study (including those withdrawn from the clinical study or lost to follow-up) shall be accounted for and documented. If a participant withdraws from the clinical investigation, the reason(s) shall be reported. If such withdrawal is due to problems related to study device safety or performance, the investigator shall ask for the participant's permission to follow his/her status/condition outside of the clinical study.

Reasons for withdrawal include:

* Physician discretion
* Participant choice to withdraw consent
* Lost to follow-up
* If the participant dies due to any cause

While study withdrawal is discouraged, participants may withdraw from the study at any time, with or without reason, and without prejudice to further treatment.

If any treated study patient is unable to return to the study center after treatment, efforts will be made to obtain complete follow-up information from the patient's primary physician. The reason for a patient's failure to return for the necessary follow-up visits or for a patient's discontinuance from the study must be determined and recorded in the case report forms (CRF).

All applicable CRFs up to the point of participant withdrawal must be completed. Participants who are "lost to follow up" should have documented attempts to contact them.

Additional data may no longer be collected after the point at which a participant has been withdrawn from the study or withdraws his/her consent, for whatever reason. Data collected up to the point of participant withdrawal may be used for study analysis.

Informed Consent All participants taking part in this clinical study must undergo the informed consent process. Participants must be allowed adequate time to review the consent, raise questions, and make a voluntary decision to participate in the clinical study. Each participant must sign and date the IRB approved informed consent form before any clinical study-related procedures are performed. A copy of signed informed consent form will be provided to the participant for his/her records. A participant's participation in the clinical study begins with the signing and dating of the informed consent form.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. At least one renal stone > 1.5 cm in maximum diameter as measured on preoperative CT scan
3. Patient is scheduled to undergo a percutaneous nephrolithotomy procedure
4. Willing and able to provide informed consent

Exclusion Criteria:

1. Pregnant
2. Active urinary tract infection
3. Prior shock wave lithotripsy within 3 months of study procedure
4. Multiple percutaneous access sites are anticipated
5. Unable or unwilling to provide informed consent -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy E Krambeck, MD, Principal Investigator — Indiana University Health
Locations (4):
- United States (3):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Indiana University Health Physicians Urology, Indianapolis, Indiana
  - The Ohio State University, Columbus, Ohio
- The University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Large T, Nottingham C, Brinkman E, Agarwal D, Ferrero A, Sourial M, Stern K, Rivera M, Knudsen B, Humphreys M, Krambeck A. Multi-Institutional Prospective Randomized Control Trial of Novel Intracorporeal Lithotripters: ShockPulse-SE vs Trilogy Trial. J Endourol. 2021 Sep;35(9):1326-1332. doi: 10.1089/end.2020.1097. Epub 2021 Aug 16. PMID 33843245

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Intention to treat - there was one patient that was recruited to the wrong arm but was maintained in that arm - and there was complete follow up with out any cross-over.
Groups:
- ShockPulse Intervention Arm: This represents patient who underwent PCNL with the ShockPulse Lithotripter
- Trilogy Intervention Arm: This represents patient who underwent PCNL with the Trilogy Lithotripter
Period: Overall Study
Arm/Group | ShockPulse Intervention Arm | Trilogy Intervention Arm
Started | 49 | 51
Completed | 49 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants of the Trilogy versus ShockPulse trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trilogy Device | ShockPulse-SE | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 49 | 100
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (14.8) | 60.4 (16.2) | 60.1 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 24 | 55
  Male | 20 | 25 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 51 | 49 | 100
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 33.4 (12.3) | 32.5 (10.1) | 32.9 (11.2)
Prior Kidney Stone Surgery [Count of Participants; unit: Participants] | 21 | 22 | 43
Surgery Study Side (Right) [Count of Participants; unit: Participants] | 23 | 23 | 46
Partial or Complete Staghorn [Count of Participants; unit: Participants] | 22 | 26 | 48
Total number of Discrete stones [Mean (Standard Deviation); unit: stones] | 2.39 (1.74) | 2.94 (2.09) | 2.67 (1.92)
Maximum Stone Diameter [Mean (Standard Deviation); unit: mm] | 23.2 (13.1) | 25.3 (10.8) | 24.3 (11)
Target Stone Hounsfield Units [Mean (Standard Deviation); unit: HU] | 927 (386) | 933 (410) | 930 (796)
Target Stone Surface Area [Mean (Standard Deviation); unit: mm^2] | 351.3 (277.7) | 375.3 (228.8) | 363.3 (114.5)
Target Stone Volume [Mean (Standard Deviation); unit: cm^3] | 4.2 (4.8) | 3.9 (3.4) | 4.1 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Stone Clearance Rate Defined as the Kidney Stone Surface Area Measured by Pre-operative Computed Tomography (CT) Scan Divided by the Time to Remove the Targeted Stone Burden.
Description: Time to remove the targeted stone burden is measured at time the lithotripter unit starts fragmenting the stone to time all fragments are removed from the kidney based on visual inspection. This is prior to final visual inspection of the kidney with a flexible nephroscope.
Time Frame: Postoperative day 1
Measure: Mean (Standard Deviation); unit: cm^3/min
Arm/Group | ShockPulse Intervention Arm | Trilogy Intervention Arm
Number analyzed (Participants) | 49 | 51
cm^3/min | 1.22 (1.67) | 0.77 (0.68)

2. Secondary Outcome: Device Malfunctions During Intraoperative Device Use as Described by Surgeon Completing the Device Questionnaire.
Description: any malfunctions during intraoperative device use
Time Frame: any malfunctions during intraoperative device use
Measure: Number; unit: malfunction events
Arm/Group | Trilogy Device | ShockPulse-SE
Number analyzed (Participants) | 51 | 49
malfunction events | 1 | 17

3. Secondary Outcome: All Complications Measured by the Clavien Classification of Surgical Complications
Description: Clavien Grade I: Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions. Acceptable therapeutic regiments are: drugs as antiemetics, antipyretics, analgetics, diuretics, electrolytes, and physiotherapy. This grade also includes wound infections opened at the bedside.
  Clavien Grade II: Requiring pharmacologic treatment with drugs other than such allowed for grade I complications. Blood transfusions and total parenteral nutrition are also included.
  Clavien Grade III: Requiring surgical, endoscopic or radiological intervention
Time Frame: 90 days
Measure: Number; unit: complications
Arm/Group | Trilogy Device | ShockPulse-SE
Number analyzed (Participants) | 51 | 49
complications
  Clavien I | 1 | 5
  Clavien II | 2 | 3
  Clavien III | 3 | 1

4. Secondary Outcome: Number of Participants With Stone Free Status as Defined by the Presence or Absence of Stone Material on Postoperative CT Imaging and at Final Follow up
Description: Stone free status must be assessed postoperative day 1 by CT scan.
Time Frame: postoperative day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Trilogy Device | ShockPulse-SE
Number analyzed (Participants) | 51 | 49
Participants | 46 | 44

ADVERSE EVENTS:
Time Frame: Monitoring of adverse events occurred throughout the trial period and 90 days after surgery.
Arm/Group | Trilogy Device | ShockPulse-SE
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/49
Other Adverse Events (participants affected / at risk) | 6/51 | 5/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trilogy Device (N=51) | ShockPulse-SE (N=49)
Hematuria (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Patient had hematuria after the procedure requiring re-admission after discharge
Hemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Hemothorax after Percutaneous Nephrolithotomy requiring chest tube placement and under anesthesia
Intesive Care Unit Admission (Infections and infestations) | 1 (1) | 1 (1) — Need for cardiopulmonary support from suspected postoperative sepsis.
Retrograde Stent Placement (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Need for additional anesthetic to replace ureteral stents after they were dislodged accidentally after surgery
Gastrointestinal Bleeding (Gastrointestinal disorders) | 1 (1) | 1 (1) — Delayed gastrointestinal bleed after Surgery requiring readmission and supportive care
Urinary Tract Infection (Infections and infestations) | 1 (1) | 2 (2) — Urinary tract infection after intervention requiring antibiotics

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT03959683/Prot_SAP_000.pdf